CLINICAL TRIAL: NCT03533517
Title: An Early Feasibility Evaluation of the AccuCinch® Ventricular Restoration System in Patients With Heart Failure and Reduced Ejection Fraction (HFrEF) - The CorCinch-HFrEF Study
Brief Title: Early Feasibility Evaluation of the AccuCinch® Ventricular Restoration System in Patients With Heart Failure and Reduced Ejection Fraction
Acronym: CorCinch-HFrEF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ancora Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 5017
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure; Cardiomyopathy, Dilated
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AccuCinch® Ventricular Restoration System (Experimental)
  Interventions: Device: AccuCinch® Ventricular Restoration

INTERVENTIONS:
Device: AccuCinch® Ventricular Restoration — AccuCinch® Ventricular Restoration System in Patients with Heart Failure and Reduced Ejection Fraction (HFrEF)

SUMMARY:
This is a non-randomized, prospective, multi-center Early Feasibility Study to evaluate the AccuCinch® Ventricular Restoration System in Patients with Heart Failure and Reduced Ejection Fraction (HFrEF).

DETAILED DESCRIPTION:
Device name changed from AccuCinch® Ventricular Repair System to AccuCinch® Ventricular Restoration System, FDA Approval Date 08Aug2020.

ELIGIBILITY:
Inclusion Criteria:

* Study patient is at least 18-years old
* Ejection Fraction: ≥20 and ≤40%
* LV end-diastolic diameter ≥55 mm
* Symptom Status: NYHA III-IV (i.e., ambulatory)
* Treatment and compliance with optimal guideline directed medical and device-based therapies for heart failure (unless contraindicated or intolerant) for at least 3 months and stable doses for 1 month with stable defined as no more than 100% increase or 50% decrease of total daily doses.
* Patients with left bundle branch block pattern and QRS duration >150ms are required to have a CRT device for at least 3 months
* Patients required to have an ICD are required to have ICD implant at least 1 month prior to enrollment
* Able and willing to complete all qualifying diagnostic and functional tests and agrees to comply with study follow-up schedule

Exclusion Criteria:

* Myocardial infarction or any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 3 months
* Mitral regurgitation grade 3 (moderate-severe) or more
* Prior surgical, transcatheter, or percutaneous mitral valve intervention
* Untreated clinically significant coronary artery disease (CAD) requiring revascularization
* Hemodynamic instability: Hypotension (systolic pressure <90 mmHg) or requirement for inotropic support or mechanical hemodynamic support
* Any planned cardiac surgery or interventions within the next 6 months (including right heart procedures)
* NYHA class IV (i.e., non-ambulatory)
* Significant RV dysfunction (TAPSE < 14)
* Severe tricuspid regurgitation
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
* Anatomical pathology or constraints preventing appropriate access/implant of the AccuCinch® Ventricular Repair System (e.g., femoral arteries will not support a 20F system)
* Renal insufficiency (i.e., eGFR of <30ml/min/1.73m2; Stage 4 or 5 CKD)
* Moderate or severe aortic valve stenosis or regurgitation or aortic valve prosthesis
* Fluoroscopic or echocardiographic evidence of severe aortic arch calcification, mobile aortic atheroma, intracardiac mass, thrombus or vegetation
* Active bacterial endocarditis
* History of any stroke within the prior 3 months or Modified Rankin Scale ≥ 4 disability from any prior stroke
* Subjects in whom anticoagulation or antiplatelet therapy is contraindicated
* Known allergy to nitinol, polyester, or polyethylene
* Any prior true anaphylactic reaction to contrast agents; defined as known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the index procedure.
* Life expectancy < 1 year due to non-cardiac conditions
* Currently participating in another interventional investigational study
* Implant or revision of any rhythm management device (CRT or CRT-D) prior 3 months or implantable cardioverter defibrillator within the prior 1 month
* Subjects on high dose steroids or immunosuppressant therapy
* Female subjects who are pregnant, of child bearing potential without a documented birth control method, or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety measured by device-related or procedure-related major adverse events (MAEs) | 30-day
  Device-related or procedure-related major adverse events (MAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, MS, CCRA, Study Director — Ancora Heart, Inc.; Ulrich Jorde, MD, Principal Investigator — Montefiore Medical Center; Azeem Latib, MD, Principal Investigator — Montefiore Medical Center
Locations (18):
- United States (18):
  - University of California, San Francisco, San Francisco, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Minneapolis Heart Foundation Institute, Minneapolis, Minnesota
  - Nebraska Heart Institute / Nebraska Heart Hospital, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mt. Sinai, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine St. Luke's Medical Center, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Carilion Roanoke Memorial, Roanoke, Virginia